CLINICAL TRIAL: NCT05995301
Title: Comparative Study on Postoperative Analgesia With Transversus Abdominis Plane Block to Local Anesthetic Infiltration With Ropivacaine in Laparoscopic Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Academy of Medical Sciences, Nepal (Other Government)
Responsible Party: Principal Investigator, Surendra Bhusal, Principal Investigator, National Academy of Medical Sciences, Nepal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NAMS Bir Hospital
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Analgesia; Ropivacaine; Laparoscopic Abdominal Surgery; Local Infiltration
Keywords: Ropivacaine; TAP Block; Analgesia; Laparoscopic abdominal surgery
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to two groups having 50patients in each, by using a computer-generated table of random numbers which was enclosed in a sealed envelope and was opened by an anesthesia assistant who was not involved in the study.
Who Masked: Participant, Care Provider
Masking Description: Patients were randomly assigned to two groups having 50patients in each, by using a computer-generated table of random numbers which was enclosed in a sealed envelope and was opened by an anesthesia assistant who was not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Transversus Abdominis Plane block
  Interventions: Drug: Ropivacaine in Transversus abdominis plane
- Group II (Experimental): Local infiltration
  Interventions: Drug: Ropivacaine in Local infiltration at port site

INTERVENTIONS:
Drug: Ropivacaine in Transversus abdominis plane — This group received 20ml of Ropivacaine 0.2% Injectable Solution in bilateral transversus abdominis plane at the end of surgery
  Arms: Group I
Drug: Ropivacaine in Local infiltration at port site — This group received local infiltration of 20ml of Ropivacaine 0.2% Injectable Solutionat port sites at the end of surgery
  Arms: Group II

SUMMARY:
The goal of this clinical trial is to compare the postoperative analgesic efficacy of ultrasound-guided TAP block with Local Anesthetic Infiltration of ropivacaine in patients undergoing laparoscopic surgery. The main question it aims to answer is:

• If Transversus Abdominis Plane block with Ropivacaine will produce long duration of analgesia than the Local Anesthetic Infiltration with ropivacaine after laparoscopic abdominal surgery .

DETAILED DESCRIPTION:
Pain is a natural phenomenon. Pain is an unpleasant sensory and emotional experience associated with actual or potential tissue damage. Pain is distressing and detrimental in post-operative patients. Management of post-operative pain has been a challenge to anesthetists. Pain treatment increase speed of recovery, minimum patient suffering, decrease length of stay, reduced hospital costs, increased patient satisfaction, increase productivity and quality of life.

Peripheral nerve blockade or field block with local anesthesia is helpful in managing postoperative pain effectively whilst avoiding complication associated with intravenous narcotics or neuraxial blockade. Regional block will help in reduction of dose and frequency of intravenous narcotics used in postoperative period, hence minimizing the side effects of narcotics.

Ultrasound guided abdominal nerve blocks are increasingly being used for anaesthesia and analgesia. The Transversus Abdominis Plane (TAP) block is a peripheral nerve block that results in anesthesia of the abdominal wall. This plane represents an anatomical potential space with nerves leaving the plane to innervate the abdominal muscles and skin. Transversus abdominis plane block (TAP block) is a novel procedure to provide postoperative analgesia following laparoscopic surgery.

Ropivacaine has a greater degree of motor sensory differentiation. Ropivacaine has been safely used up to the dose of 200 mg (100 ml of 0.2% ropivacaine) as a field block for post operative analgesia. We are giving a larger volume of ropivacaine (20 ml on each side) expecting to cover the upper abdomen when TAP block is performed via posterior approach.

NULL HYPOTHESIS There is no difference in post operative analgesia with Transversus Abdominis Plane block and local anesthetic infiltration after laparoscopicabdominal surgery

General objective

1. To compare the efficacy of Transversus Abdominal plane block and local anesthetic infiltration after laparoscopic abdominal surgery

Specific objective

1. To compare the visual analog score (VAS) between two groups
2. To compare time to first analgesic requirement between two groups.
3. To compare the total dose of analgesia in 24 hours between the two groups

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of either sex aged 25-70 years
2. ASA physical status I or II
3. Patient posted for elective abdominal laparoscopic surgery.

Exclusion Criteria:

1. Any absolute contraindications to peripheral nerve blockade
2. History of Hypersensitivity to Drugs
3. Uncontrolled Diabetes Mellitus, Renal Failure, Hepatic failure
4. History of neuromuscular or psychiatric disease
5. Patient receiving psychotropic drug, chronic analgesic therapy
6. Pregnancy
7. Patient weight less than 50 kg

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | Time Frame: upto first 24 hour after intervention
  Visual analog scale at rest

SECONDARY OUTCOMES:
Duration of analgesia | Time Frame: upto first 24 hour after intervention
  Visual analog scale on movement

OTHER OUTCOMES:
Time to first rescue analgesia | Time Frame: upto first 24 hour after intervention
  The time of first complaint of pain by the patient.
Total pethidine consumption | Time Frame: upto first 24 hour after intervention
  At any point of time when VAS was>3, injection pethidine 0.5 mg/kg and injection promethazine 0.25 mg/kg was given via intravenous route
Total ketorolac consumption | Time Frame: upto first 24 hour after intervention
  When pain persisted for more than 15 min after giving intravenous pethidine, injection ketorolac 30 mg intravenous was given

CONTACTS AND LOCATIONS:
Overall Officials: Surendra Bhusal, MD, Principal Investigator — NAMS Bir Hospital; Brihaspati K C, MD, Study Director — NAMS Bir Hospital; Kaushal Tamang, MD, Study Chair — NAMS Bir Hospital
Locations (1):
- National Academy of Medical Sciences, Kathmandu, Bagmati, Nepal